CLINICAL TRIAL: NCT04988919
Title: Acute Consumption of 4D Dietary Supplement vs. Placebo: Effects on Perceptual-Cognitive and Visual-Motor Performance
Brief Title: Consumption of 4D Dietary Supplement on Perceptual-Cognitive and Visual-Motor Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Collaborators: 4D, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: STUDY00003029
Record Dates: First submitted 2021-07-14; First posted 2021-08-04 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Dietary Supplementation
Keywords: multi-ingredient supplement; reaction time; reactive agility; cognition

STUDY DESIGN:
Intervention Model Description: Participants will consume the 4D dietary supplement and the placebo in a randomized order on different testing days. Both the supplement and the placebo will be mixed with 24 fluid ounces of water. All drinks will have a similar appearance and taste. Researchers and participants will be blinded to the contents.
Who Masked: Participant, Investigator
Masking Description: All investigators and participants will be blinded to the treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4D dietary supplement (Experimental): Multi-ingredient supplement containing a proprietary blend with 150mg of caffeine, and other ingredients including vitamins, electrolytes, and BCAA blend (150mg).
  Interventions: Dietary Supplement: 4D
- placebo (Placebo Comparator): flavored water (raspberry lemonade Crystal Light®)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: 4D — multi-ingredient supplement mixed with 24 ounces of water
  Arms: 4D dietary supplement
Dietary Supplement: placebo — taste-matched placebo mixed with 24 ounces of water
  Other Names: Crystal Light®
  Arms: placebo

SUMMARY:
The purpose of this investigation is to determine if supplementation with the 4D dietary supplement impacts perceptual-cognitive and visual-motor skills in healthy individuals.

DETAILED DESCRIPTION:
Multi-ingredient supplements (MIS) have been reported to positively impact various aspects of performance. While caffeine alone has been shown to improve aerobic performance, resistance training (such as bench press), reaction time and sprint performance, it has also been suggested that it lacks the ability to improve cognition. Therefore, the purpose of this investigation is to examine the effects of a caffeine containing MIS on measures of cognition and reaction time, with the intent of providing additional benefits to athletic performance.

This study will utilize a randomized, double-blind, placebo-controlled design. Following two familiarization trials, participants will complete two testing visits. During these visits, they will complete baseline assessments, consume either the 4D dietary supplement or a taste matched placebo, and rest for 45 minutes. Reaction time, cognition assessments (visual tracking speed), and reactive agility performance will be assessed following the rest period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 18-40 years old
* Determined to be healthy by the MHQ and PAR-Q+

Exclusion Criteria:

* Any response of "yes" on the PAR-Q+
* Daily caffeine consumption greater than 200 mg

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Change in reactive agility time | post supplement ingestion on both testing days (Day 3 and Day 4)
  Determined via Y-Reactive Agility test using the Witty Wireless Timing Gate system
Change in reaction time in response to supplement/placebo consumption | pre and post supplement ingestion on both testing days (Day 3 and Day 4)
  Determined via Dynavision D2, Mode A
Change in visual tracking speed in response to supplement/placebo consumption | pre and post supplement ingestion on both testing days (Day 3 and Day 4)
  Determined via multiple object tracking test on the Neurotracker

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Florida, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No